CLINICAL TRIAL: NCT03348501
Title: Study and Follow-up of Multiple Endocrine Neoplasia Type 1
Acronym: GENEM
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GOUDET PARI2011
Record Dates: First submitted 2017-11-13; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Multiple Endocrine Neoplasia
MeSH Terms: conditions — Multiple Endocrine Neoplasia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum 6 ml of blood and tissue 50 mg of tumour
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey for long-term follow-up of the disease — patients will be regularly asked about their state of health (occurrence of a major health event that required hospitalization, for example ...), and about their living conditions (alcohol and tobacco consumption, socio-economic environment). Questionnaires of quality of life and satisfaction related to care will also be offered at regular intervals to better know the impact of their disease on their daily lives and their perception of their care.

SUMMARY:
Multiple Endocrine Neoplasia type I (MEN1) or Wermer syndrome is an autosomal dominant disease that predisposes patients to the development of endocrine tumours, principally parathyroid, pituitary or duodenal-pancreatic tumours. It is due to mutations that abolish the function of the MEN1 gene, which contributes to tumour regulation. It is a rare disease, with an estimated prevalence in the general population of 1/30,000. Penetrance of the disease is late but very high (almost 100% at 50 years of age). The first clinical manifestations usually appear after the age of 30 or 40 years.

The three cardinal endocrine characteristics of MEN1 are secreting tumours of the parathyroid, the pituitary gland and the pancreas. Tumours of the adrenal glands, bronchial or thymic endocrine tumours, ependymoma and meningioma of the central nervous system, visceral leiomyomas, and certain cutaneous tumours can also be found as well as these cardinal tumours.

The diagnosis of MEN1 is essential to ensure 1) appropriate therapeutic management of the proven endocrine manifestations 2) screening for other endocrine and non-endocrine tumours (lesions), 3) family screening of affected relatives whether they are symptomatic or not 4) the surveillance of thus diagnosed patients. Studies on mortality in MEN1 have shown that the causes of death are mainly due to the disease. The non-diagnosis of MEN1 is a cause of therapeutic failure in the management of the endocrine lesions. For the success of the surgical treatment of an isolated endocrine lesion it is important for patients to be oriented towards a diagnosis of MEN1 as the management is different from that in usual situations. Detection is thus of major importance, as early diagnosis can improve the management.

Even though the syndrome was discovered in 1903 by Erdheim and correctly documented in 1954 by Wermer, it was only in the 1970s that we became aware of the variety of clinical forms and attempted to codify its treatment. Nonetheless, published studies are fragmented and concern selected populations of few patients. They only partially answer questions arising in clinical practice concerning the prognosis and optimal management of patients. The natural history of the disease in all of its clinical forms is still poorly understood. Although advances in genetics have helped in the diagnosis of MEN1, some clinical forms are still difficult to associate with the syndrome: atypical forms, forms with hardly any symptoms and no genetic diagnosis (10%). These clinical forms need to be clarified to ensure optimal care. Only a large cohort will make it possible to describe the different forms of this disease and to clarify its prognosis

ELIGIBILITY:
Inclusion Criteria:

- Symptomatic individuals with a confirmed diagnosis of MEN1 and who live in France.

Patients with the following characteristics will also be included in the cohort:

* At least two of the three cardinal clinical lesions (parathyroid, pancreas, pituitary),
* OR an isolated known lesion of the disease, cardinal or not (parathyroid, pancreas, pituitary, adrenal, thymus, bronchus, tumour of the central nervous system) associated with a mutation of the MEN1 locus on chromosome 11q13,
* OR an isolated lesion, cardinal or not (parathyroid, pancreas, pituitary, adrenal, thymus, bronchus, tumour of the central nervous system) in an individual with a confirmed family history of MEN1.

asymptomatic patients who carry a characteristic mutation of MEN1. Current knowledge suggests that these patients will develop symptoms during their follow-up.

Exclusion Criteria:

patients who present a single-organ genetic endocrine disease associated with another genetic syndrome (familial isolated pituitary adenoma FIPA, familial isolated hyperparathyroidism FIHP)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This cohort includes symptomatic individuals, whose diagnosis of NEM1 has been confirmed, and domiciled in France
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Questionnaire or Life quality | through study completion, an average of 19 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France